## PRINCIPAL INVESTIGATOR: Christian Hinrichs, MD

STUDY TITLE: A Phase II Study of Immunotherapy with E7 T Cell Receptor T Cells for

Vulvar High-Grade Squamous Intraepithelial Lesions

**STUDY SITE: NIH Clinical Center** 

Cohort: Treatment

Consent Version: 4/27/2020

# WHO DO YOU CONTACT ABOUT THIS STUDY?

**Principal Investigator:** Christian Hinrichs, MD

Phone: 240-760-6059 Email: <u>Hinrichs@nih.gov</u>

## KEY INFORMATION ABOUT THIS RESEARCH

This consent form describes the research study and is designed to help you decide if you would like to be a part of the research study.

You are being asked to take part in a research study at the National Institutes of Health (NIH). This section provides the information we believe is most helpful and important to you to in making your decision about participating in this study. Additional information that may help you make a decision can be found in other sections of the document. Taking part in research at the NIH is your choice.

You are being asked to consider joining this study because you have been diagnosed with a human papillomavirus (HPV)-16 associated premalignant condition of the vulva (high-grade squamous intraepithelial lesion (HSIL).

The purpose of this research study is to determine if a personalized immune treatment can rid the body of HPV infection and thereby cure vulvar HSIL.

If you decide to join this study, here are some of the most important things that you should know that will happen:

- You may only participate in this study if you have vulvar HSIL that cannot be removed with surgery without causing disfigurement or functional impairment that you would consider unacceptable, or if you have already had surgery but it failed to control your vulvar HSIL.
- The primary treatment is surgery to cut out the areas of HSIL. Sometimes a cream that stimulates the immune system may also be used for treatment. Rarely, vulvar HSIL can go away on its own.
- The therapy used in this study is called T cell therapy. Immune cells from your blood will be genetically modified in the laboratory to give them the ability to attack the human papillomavirus.

## PATIENT IDENTIFICATION

- Screening tests are required prior to you receiving the study drug. If you are found eligible for the study, you will undergo a procedure to collect your T cells from the peripheral blood. These cells will be modified in the laboratory and will be given back to you by a one-time infusion into a vein. You will stay in the hospital for 1-2 days.
- You may experience side effects from taking part in this study. Most are likely to be mild which may include fever or chills. It is possible that you could develop more serious, temporary, long-lasting or permanent side effects including death.
- You will be seen regularly during the study. You will have clinical, laboratory and imaging tests to done to see how you are doing and to assess your disease. We will also collect required samples from you including biopsies of your disease and blood samples for both clinical and research purposes.
- After the study follow-up period has ended, we would like to talk with you once a year for 5 years from the day of treatment to see how you are doing. We will ask you to participate in a long term follow-up study where we will follow you for 15 years from the time you receive the cells.

Just as we do not know what side effects you might have, we cannot know if you may benefit from taking part in this study. If you do not benefit, this study and the results from our research may help others in the future.

The remaining document will now describe this research study in more detail. This information should be considered before you make your choice. Members of the study team will talk with you about all the information described in this document. Some people have personal, religious, or ethical beliefs that may limit the kinds of medical or research treatments they would want to receive (such as blood transfusions). Take the time needed to ask any questions and discuss this study with NIH staff, and with your family, friends, and personal health care providers.

If the individual being asked to participate in this research study is not be able to give consent to be in this study, you are being asked to give permission for this person as their decision-maker. The term "you" refers to you as the decision-maker and/or the individual being asked to participate in this research, throughout the remainder of this document.

## IT IS YOUR CHOICE TO TAKE PART IN THE STUDY

You may choose not to take part in this study for any reason. If you join this study, you may change your mind and stop participating in the study at any time and for any reason. In either case, you will not lose any benefits to which you are otherwise entitled. However, to receive care at the NIH, you must be taking part in a study or are being considered for a study. If you do choose to leave the study, please inform your study team to ensure a safe withdrawal from the research.

#### WHY THIS STUDY IS BEING DONE?

This is a research study. We are investigating an experimental therapy with genetically modified immune cells that target the human papillomavirus (HPV) for vulvar high-grade squamous intraepithelial lesion (HSIL). Vulvar HSIL is caused by infection of the vulva with HPV. In a small percent of patients vulvar HSIL can turn into cancer. The risk of cancer can be reduced by

NIH-2977 (4-17)


File in Section 4: Protocol Consent (1)

Version Date: 4/27/2020

IRB NUMBER: 19C0091

NIH) IRB APPROVAL DATE: 06/04/2020

treatment of HSIL. The primary treatment is surgery to cut out the areas of HSIL. Sometimes a cream that stimulates the immune system may also be used for treatment. Rarely, vulvar HSIL can go away on its own.

Surgery for vulvar HSIL can cause disfigurement or functional impairment. Also, it may not completely remove the disease and may not prevent its recurrence. You may only participate in this study if you have vulvar HSIL that cannot be removed with surgery without causing disfigurement or functional impairment that you would consider unacceptable, or if you have already had surgery but it failed to control your vulvar HSIL.

The purpose of this research study is to determine if a personalized immune treatment can rid the body of HPV infection and make your HSIL lesions go away. The immune treatment in this study is called T cell therapy. Immune cells from your blood will be genetically modified in the laboratory. The genetically modified cells will then be given back to you through an intravenous infusion similar to a blood transfusion.

In this study we are modifying your immune cells with a retrovirus to give them the ability to attack HPV-16 E7, a protein that is part of HPV. The HPV-16 E7 protein has been found only on cells infected with the HPV virus. We have given immune cells modified with the same genes to other patients. Our laboratory studies show that these cells work much like the cells we have given patients in the past and should be just as safe as those cells, however, we can't predict all of the side effects that may occur.

In a previous clinical trial with E7 TCR T cells, patients had metastatic HPV16+ cancers. Different amounts of cells were given to these patients. The cell infusions were well-tolerated. Tumor responses occurred in 6 of 12 patients; responses were seen at all dose level of cells. In that trial, patients received chemotherapy prior to cell infusion followed by aldesleukin, which is thought to increase both the clinical activity and the toxicity of the T cells. In the current trial, patients will not receive chemotherapy or aldesleukin.

We are asking you to join this research study because you have been diagnosed with an HPV-16 associated premalignant condition of the vulva (high-grade squamous intraepithelial lesion (HSIL). In addition, you completed the screening evaluation and were found to be eligible to participate in this research study.

E7 TCR T cells are considered investigational, which means that it has not been approved by the U.S. Food and Drug Administration (FDA) to treat vulvar HSIL.

# WHAT WILL HAPPEN DURING THE STUDY?

The cell therapy protocol has several stages that happen after screening is complete. These are listed below:

| Stage | Timeframe | Location | Comments & Instructions |
|---|---|---|---|
| Baseline testing | Occurs over 1-2<br>weeks | Outpatient | Optional vulvar biopsy, photographs of lesion(s), labs, other tests as needed |
| Leukapheresis | Occurs on one | Outpatient | This is a half to full day appointment. |

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 4/27/2020


| (see page 4 of<br>this consent<br>document) | day, at least 21<br>days prior to cell<br>infusion | | |
|---|---|---|---|
| Cells (Day 0) | 1 day | Inpatient | Receive the E7 TCR cells IV |
| Recovery | 1-3 days | Inpatient unit | Recover from the effects of treatment. |
| Protocol<br>Follow-up | Ongoing for up to 2 years. | Outpatient | Return to NIH clinic for physical exam, review of side effects, labs |
| Local<br>Follow-up | Annually for years 3-5 | Outpatient | Annual history and physical exam from a healthcare provider (may be performed outside NIH) |
| Long-term follow-up | Annually for years 6-15 | Phone/mail | Answer questionnaire via telephone or mail |

# **During the study**

# Cell harvest and growth

You will undergo leukapheresis to obtain your white blood cells. These cells will be grown in the lab and genetically modified to recognize a protein on your precancerous cells. If your cells do not grow, you will not be able to receive the cell infusion. If that happens, we will look at alternative experimental treatments at the NIH Clinical Center or refer you to the care of your referring physician. We usually know after about 4 weeks whether the cells will grow well enough to be used as an experimental treatment on this protocol. At the time we determine that your cells are not growing, we will inform you and discuss your options with you. If you were previously treated on protocol 17-C-0116, your cell product will be made from cells that were collected while you were treated on that protocol.

# Leukapheresis

Leukapheresis is a procedure that allows us to remove certain types of blood cells from you and return the rest of your blood. It is a very common procedure that is done routinely here at the NIH with very few risks. During leukapheresis, blood is removed from you through a needle in your arm, circulated through a machine that divides whole blood into red cells, plasma (the serum part), and leukocytes (or white cells), and then the plasma and red cells are returned to you through a second needle in your other arm. If you are receiving the experimental cell therapy, the white blood cells will be used to grow your treatment cells. In addition to the leukapheresis you will undergo as part of your work up, we will also ask you to undergo one additional pheresis procedure for the purpose of research between 4 and 6 weeks after your cell treatment to see the impact of this therapy on the immune system and see if cells we gave you are still active. If you were previously treated on protocol 17-C-0116, you will only undergo a single leukapheresis procedure between 4 and 6 weeks.

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)


File in Section 4: Protocol Consent (1)

Version Date: 4/27/2020

# Cell Infusion (Day 0)

You will be admitted to the hospital for this procedure. You will be given the cells through an IV (intravenously, or through your veins) over 20 to 30 minutes on day 0. This may be done through a peripheral line (a short tube placed in a vein in your arm), through a "central line," (an IV catheter [or tube] placed in the large vein in your neck or in your chest, or through a PICC line (a peripherally inserted central catheter, which is a thin tube inserted into a vein in your upper arm and is then guided into a large vein in your chest). The doctor will discuss this with you to determine the best method for you. The day after your cells are infused, we will watch you closely during this entire time for any side effects of this experimental regimen. We will discuss the side effects below and we will include in your care all the medicines and treatments to prevent as many of these side effects as we can and to make you as comfortable as we can.

# When you are finished with the T cell treatment

## Recovery

You will recover in the hospital until you are well enough to go home. This usually takes 1-3 days after you have received cells; however, you may need to stay in the hospital for longer than this before you are well enough to go home. We will continue to give you support medications, do laboratory tests, and watch you closely for any side effects until we feel your condition is stable.

In addition to the laboratory tests to monitor your condition, we will remove between 1 and 9 teaspoons of blood for research one day after you have received cells, three days after you have received cells, then three days per week for one week (Monday, Wednesday, Friday) and then once per week until you are discharged from the hospital to study the effects of this regimen on your immune system. If you experience side effects in your kidneys, we will collect 1 additional teaspoon of blood and about 6 teaspoons of urine to help us determine the cause of these side effects. The maximum amount of blood for research is approximately 2.3 cups in 8 weeks.

# Follow up and Evaluation of Experimental Regimen

We will ask you to return to the NIH Clinical Center frequently for follow-up visits after you are discharged approximately every month for 3 months. After 3 months, if your lesions have not shrunk, you will need to follow up with your physician for care. If your lesions have shrunk after 3 months, you will be seen monthly for another 3 months. If at 6 months, your lesions are still present, you will need to follow up with your physician for care. If at 6 months, your tumor has disappeared, you will be seen every three months for two visits, then every 6 months for 2 visits. The follow up visits will probably take about 1 day. At each visit, you will have lab tests and a physical examination. At some of your follow up visits, you may undergo leukapheresis or have about 8 tubes of blood drawn (4 tablespoons) for research so that we can see the effect this therapy has had on your immune system and if the cells we gave you are still alive. At some follow-up visits you will have a vulvar biopsy performed (at your 2-week follow-up, your 1-month follow-up visit, and at the last follow-up visit). There will be a separate consent for any biopsies.

## PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17)

Once you are done with your regular visits, we will contact you or your physician once a year for five years after your last dose of cell therapy to ask you questions about your HSIL, such as whether you have had procedures or other treatments.

#### Retreatment

If your HSIL shrank or disappeared following the initial treatment, you may be able to receive one additional treatment of E7 TCR T cells if you tolerated the first treatment well. You will receive the same cell infusion on the same schedule as with the first treatment. You will be allowed to have the second treatment only if we have enough of your cells left over from the first treatment you had. The study doctors will review this with you. The second treatment will not begin until at least 12 weeks after your first treatment. Gene Therapy Long Term Follow up (Retroviral Vectors)

Because we do not know the long-term side effects of gene therapy, we will collect your blood over the next several years, frequently at first and then less frequently. We can obtain the blood needed for these studies at your regular follow-up visits as long as you are on the study. If you are removed from the study, we still need to conduct these gene-therapy follow-up visits according to FDA regulations and will request your permission to enroll you in a protocol that would allow us to follow you for this reason only. If you return to your referring physician after receiving therapy here, we will ask you to have your physician send your blood specimens here for this testing, which will decrease the inconvenience to you. This testing will determine if the cells have grown or changed in your body. We will test your blood immediately before you receive the cells, and then at 3, 6, and 12 months. If all the tests are normal and show no change, we will collect blood from you every year after that to store in case you develop symptoms later. According to FDA requirements, you need to have an annual physical examination at the NIH or with your local provider for five years after you receive the cells. After that time, we will be sending you a questionnaire to get information regarding your health for the next ten years, for a total follow-up time period of 15 years. For this reason, we ask that you continue to provide us with a current address and telephone number, even after you complete this research study. At the time of your death, no matter the cause, we may request permission for an autopsy to obtain vital information concerning the safety of this experimental therapy approach. Please discuss this request with your family to inform them of your wishes.

## HOW LONG WILL THE STUDY TAKE?

If you agree to take part in this study, your involvement will last for up to 5-years:

- You may be seen in the clinic for 5 times in the first 3 months after receiving E7 T cells. The rest of the follow-up visits will depend on if your disease is growing.
- If after 3 months your disease is not getting smaller or it is growing, then you will need to follow up with your gynecologist at home for further treatment options. We will contact you once a year to ask you questions about your disease and any treatments for the disease that you have received. This will happen for a total of 5 years.

Your involvement on the Gene Therapy Long Term Follow Up Study will be 15 years once you receive the E7 T cells on this study. The FDA requires an annual physical exam with a healthcare

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


provider at or outside the NIH for five years after receiving the E7 T cells, followed by annual phone or mail questionnaire until 15 years after receiving the E7 T cells.

## HOW MANY PEOPLE WILL PARTICIPATE IN THIS STUDY?

Approximately 16 people will participate in this study at the NIH.

# WHAT ARE THE RISKS AND DISCOMFORTS OF BEING IN THE STUDY?

# What side effects or risks can I expect from the study therapy and procedures?

The risks and discomforts of this research study can be significant. It is possible, although unlikely, that this experimental treatment may cause your death.

We will discuss the side effects of this experimental treatment with you. You will be given medicines, transfusions, and treatments as needed to prevent or treat the side effects. We will try to make you as comfortable as possible.

# Leukapheresis

During the leukapheresis procedure, you may have some tingling in your face and lips due to the medicine used to keep your blood from clotting during the procedure. The nurses may give you a calcium-containing antacid to chew that takes away this tingling. Rarely, people may experience lightheadedness or dizziness. We ask that you eat prior to the procedure to prevent this. Rare complications of this procedure are lowered blood pressure, bleeding or bruising where the needles are put in your arms.

## **Cell Infusion**

The cells we will be giving you have a type of virus (retrovirus) put into them that makes them able to recognize the HPV E7 protein. Although this retrovirus is not active, there is the rare possibility that it may cause infection. The cells could also cause you to develop another type of cancer, such as leukemia or lymphoma.

Potential risks include:

- Fever, chills and shortness of breath, which may last for a few hours (common)
- Lung congestion causing shortness of breath
- Severe reaction to the cells which would include very low blood pressure and damage to your heart, lung, and/or kidneys
- As this is a new experimental therapy which has not been given to patients with your disease, side effects that we do not anticipate that may cause your condition to deteriorate may be encountered. Any new information that becomes available during the course of this study will be shared with you.

# **Intravenous Line Placement**

You will require either a peripheral or central line catheter. If you require a peripheral IV line, the risks include pain, bleeding, infection and rash/swelling at the insertion site.

Insertion of a peripherally inserted central catheter (PICC) may require local anesthesia. PICC lines enter the body through the skin usually in the arm and extend to the heart. The risks of the

# PATIENT IDENTIFICATION


insertion procedure include pain, bleeding, rash/swelling at the insertion site and infection. Long-term risks of a PICC line include infection, a blockage from air that gets into a vein, or a blood clot in the vein. If these occur, it may be necessary to remove the PICC line. These risks will be explained to you in more detail at the time of insertion.

If you require a Central line catheter, it is usually inserted under local anesthesia. The risks associated with the procedure include pain, bleeding, infection, and puncture of the underlying lung. Lung puncture can result in lung collapse, which might require that a chest tube be placed into the chest cavity (usually for a day or two) to help the lung re-inflate. The long-term risks of the catheter include infection and clotting of the vein in which the catheter sits. If these occur, it may be necessary to remove the catheter. These risks will be explained to you in more detail at the time of the insertion.

# Optional vulvar biopsy risks

The risks of a vulvar biopsy include bruising and discomfort at the biopsy site and rarely bleeding and infection.

Prior to and throughout this study you will undergo many physical exams to determine the size and extent of your precancer lesion, as well as the impact of the treatment. Multiple blood tests will be performed and some of your serum and lymphocytes will be stored for future testing. Blood and tissue samples collected from you may be stored and used in the future to study scientific questions related to this protocol. If there are any risks to you or your family associated with these future scientific studies which are not covered in this consent form, your consent will be obtained before such studies are performed.

If your disease progresses or recurs after this experimental treatment, then you will no longer receive treatment in this protocol, though you may be eligible to be considered for other protocols at the National Cancer Institute, NIH or referred elsewhere for treatment.

# Gene Therapy Risk of Cancer and Other Diseases

We are unsure if this type of gene therapy will cause you to become sick in the future. It is possible that it may cause your immune system or nerves not to work well or cause a sickness of your blood cells or even a cancer (for example leukemia). We do not know if you will develop any of these disorders, but you need to be aware of this possible risk. Children in France and England received gene therapy for a particular disease of the immune system. Most of the children were cured, but 5 children out of 22 later developed leukemia and one died. Experts who looked at these cases thought that the gene therapy caused the leukemia in these children. To watch you for this risk we will be testing your blood as described before.

You will be treated on this gene transfer protocol with a viral vector that was manufactured at the NCI Surgery Branch Vector Production Facility before May 2016. An internal review of the facility that made the vector for this protocol determined that the facility needed to be closed due to manufacturing issues. We know of no additional risks related to the previously produced vector for patients who have received cells with vectors made in this facility as the vectors were extensively tested by outside experts. Therefore, the IRB has determined that the potential benefit to you outweighs the potential risks.

# **Blood Draws**

## PATIENT IDENTIFICATION

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)




Blood will be drawn frequently during your treatment. Most of the blood draws will be to monitor your health during and after the T-cell infusion. In addition, some blood samples will be drawn for research purposes. Additional blood draws might be necessary to investigate T cell responses and serum cytokine levels in cases of clinical events such as rapid regressions of lesions or toxicity. These samples will be used to study how your immune system is affected by the cell therapy. Some of the samples may be used for other or future research conducted by the investigational team or other researchers. Side effects of repeated blood sampling depend in part on how the blood is drawn. If through a central venous catheter, risks include contamination of the catheter which would result in a serious blood stream infection, requiring admission to the hospital and giving you antibiotics through the vein; if blood is drawn through a needle into your skin, side-effects could include pain and bruising in the area where the blood was drawn. Other side-effects can include lightheadedness, or rarely, fainting. If you have too much blood taken over a prolonged period, your red blood cell count may drop (this is called "anemia"). As a precaution, we will check your red blood cell level, and give you iron treatment or a blood transfusion if needed.

# What are the risks related to pregnancy?

If you are able to become pregnant, we will ask you to have a pregnancy test before starting this study. You will need to practice an effective form of birth control before starting study treatment, during study treatment, and for 4 months after you finish study treatment (the restricted period). If you become pregnant, there may be unknown risks to the fetus or unborn child, or risks that we did not anticipate. There may be long-term effects of the treatment being studied that could increase the risk of harm to a fetus. You must tell the study doctor if your birth control method fails during the restricted period. If you think or know you have become pregnant during the restricted period, please contact the study team as soon as possible. Please discuss with the research team how long you need to wait before becoming pregnant after completing the course of this study drug or procedures on this study.

You may not participate in this study if you are pregnant. If you are capable of becoming pregnant, we will perform a pregnancy test before exposing you to radiation. You must tell us if you may have become pregnant within the previous 14 days because the pregnancy test is unreliable during that time.

## WHAT ARE THE BENEFITS OF BEING IN THE STUDY?

You might not benefit from being in this study.

However, the potential benefits could include shrinking of your precancer or lessening of your symptoms, such as pain, that are caused by the lesions.

# Are there any potential benefits to others that might result from research?

In the future, other people might benefit from this study because the knowledge gained from this study may help in developing treatments for those who have this precancer.

## WHAT OTHER OPTIONS ARE THERE FOR YOU?

Before you decide whether or not to be in this study, we will discuss the other options that are available to you. Instead of being in this study, you could:

#### PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 4/27/2020


- Get treatment or care for your precancer without being in a study, such as surgery to remove the lesion(s). This is called surgical excision. Another treatment option for some individuals is topical imiguimod, a cream that is applied directly to the lesions.
- Take part in another study

Please talk to your doctor about these and other options.

#### DISCUSSION OF FINDINGS

# New information about the study

If we find out any new information that may affect your choice to participate in this study, we will get in touch with you to explain what we have learned. This may be information we have learned while doing this study here at the NIH or information we have learned from other scientists doing similar research in other places.

#### Return of research results

We do not plan to return research results to you. A summary of the research results will be posted on Clinicaltrials.gov at completion of the study.

## EARLY WITHDRAWAL FROM THE STUDY

Your doctor may decide to stop your therapy for the following reasons:

- if he/she believes that it is in your best interest
- if you become pregnant
- if your disease comes back during treatment
- if you have side effects from the treatment that your doctor thinks are too severe
- if the sponsor, the FDA, the Institutional Review Board or your doctor decides to stop or interrupt the study
- if new information shows that another treatment would be better for you

In this case, you will be informed of the reason therapy is being stopped.

You can stop taking part in the study at any time. However, if you decide to stop taking part in the study, we would like you to talk to the study doctor and your regular doctor first.

If you decide at any time to withdraw your consent to participate in the trial, we will not collect any additional medical information about you. However, according to FDA guidelines, information collected on you up to that point may still be provided to our collaborators or their designated representatives.

# STORAGE, SHARING AND FUTURE RESEARCH USING YOUR SPECIMENS AND **DATA**

## Will Your Specimens or Data Be Saved for Use in Other Research Studies?

As part of this study, we are obtaining specimens and data from you. We will remove all the identifiers, such as your name, date of birth, address, or medical record number and label your

specimens and data with a code so that you cannot easily be identified. However, the code will be linked through a key to information that can identify you. We plan to store and use these specimens and data for studies other than the ones described in this consent form that are going on right now, as well as studies that may be conducted in the future. These studies may provide additional information that will be helpful in understanding vulvar HSIL, or other diseases or conditions. This could include studies to develop other research tests, treatments, drugs, or devices, that may lead to the development of a commercial product by the NIH and/or its research or commercial partners. There are no plans to provide financial compensation to you if this happens. Also, it is unlikely that we will learn anything from these studies that may directly benefit you.

I give permission for my coded specimens and data to be stored and used for future research as described above.

| Yes | No |
|----------|----------|
| Initials | Initials |

# Will Your Specimens or Data Be Shared for Use in Other Research Studies?

We may share your coded specimens and data with other researchers. If we do, while we will maintain the code key, we will not share it, so the other researchers will not be able to identify you. They may be doing research in areas similar to this research or in other unrelated areas. These researchers may be at NIH, other research centers and institutions, or industry sponsors of research.

I give permission for my coded specimens and data to be shared with other researchers and used by these researchers for future research as described above.

| Yes | No |
|----------|----------|
| Initials | Initials |

If you change your mind and do not want us to store and use your specimens and data for future research, you should contact the research team member identified at the top of this document. We will do our best to comply with your request but cannot guarantee that we will always be able to destroy your samples. For example, if some research with your specimens and data has already been completed, the information from that research may still be used. Also, if the specimens and data have been shared already with other researchers, it might not be possible to withdraw.

In addition to the planned use and sharing described above, we might remove all identifiers and codes from your specimens and data and use or share them with other researchers for future research at the NIH or other places. When we or the other researchers access your anonymized data, there will be no way to link the specimens or data back to you. We will not contact you to ask your permission or otherwise inform you before we do this. We might do this even if

## PATIENT IDENTIFICATION

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)


you answered "no" to the above questions. If we do this, we would not be able to remove your specimens or data to prevent their use in future research studies, even if you asked, because we will not be able to tell which are your specimens or data.

NIH policies require that your clinical and other study data be placed in an internal NIH database that is accessible to other NIH researchers for future research. These researchers will not have access to any of your identifiers, such as your name, date of birth, address, or medical record number; and your data will be labeled with only a code. We cannot offer you a choice of whether your data to be placed in this database or not. If you do not wish to have your data placed in this database, you should not enroll in this study.

# How Long Will Your Specimens and Data be Stored by the NIH?

Your specimens and data will be stored at NIH indefinitely.

# Risks of Storage and Sharing of Specimens and Data

When we store your specimens and data, we take precautions to protect your information from others that should not have access to it. When we share your specimens and data, we will do everything we can to protect your identity by removing information that can identify you. Even with the safeguards we put in place, we cannot guarantee that your identity will never become known or someone may gain unauthorized access to your information. New methods may be created in the future that could make it possible to re-identify your data or specimens.

# COMPENSATION, REIMBURSEMENT, AND PAYMENT

# Will you receive compensation for participation in the study?

Some NIH Clinical Center studies offer compensation for participation in research. The amount of compensation, if any, is guided by NIH policies and guidelines.

You will not receive compensation for participation in this study.

# Will you receive reimbursement or direct payment by NIH as part of your participation?

Some NIH Clinical Center studies offer reimbursement or payment for travel, lodging or meals while participating in the research. The amount, if any, is guided by NIH policies and guidelines.

On this study, the NCI will cover the cost for some of your expenses. Some of these costs may be paid directly by the NIH and some may be reimbursed after you have paid. Someone will work with you to provide more information.

# Will taking part in this research study cost you anything?

NIH does not bill health insurance companies or participants for any research or clinical care that you receive at the NIH Clinical Center.

- If some tests and procedures are performed outside the NIH Clinical Center, you may have to pay for these costs if they are not covered by your insurance company.
- Medicines that are not part of the study treatment will not be provided or paid for by the NIH Clinical Center.

## PATIENT IDENTIFICATION

 Once you have completed taking part in the study, medical care will no longer be provided by the NIH Clinical Center.

# **CONFLICT OF INTEREST**

The National Institutes of Health (NIH) reviews NIH staff researchers at least yearly for conflicts of interest. This process is detailed in a COI Guide. You may ask your research team for a copy of the COI Guide or for more information. Members of the research team who do not work for NIH are expected to follow these guidelines or the guidelines of their home institution, but they do not need to report their personal finances to the NIH.

The National Institutes of Health and the research team for this study are using E7 TCR (biological product) developed by Center for Cancer Research through a joint study with your study team and Kite Pharma. This means it is possible that the results of this study could lead to payments to NIH. By law, the government is required to share such payments with the employee inventors. You will not receive any money from the development of E7 TCR.

Kite Pharma will provide financial support for this study.

# CLINICAL TRIAL REGISTRATION AND RESULTS REPORTING

A description of this clinical trial will be available on <a href="http://www.clinicaltrials.gov">http://www.clinicaltrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

# CONFIDENTIALITY PROTECTIONS PROVIDED IN THIS STUDY

Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database. Your test results will be identified by a unique code and the list that links the code to your name will be kept separate from your sample and health information. Your information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like tuberculosis. However, the researchers will do their best to make sure that any information that is released will not identify you.

# Will your medical information be kept private?

We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Organizations that may look at and/or copy your medical records for research, quality assurance, and data analysis include:

- The NIH and other government agencies, like the Food and Drug Administration (FDA), which are involved in keeping research safe for people.
- National Institutes of Health Intramural Institutional Review Board
- The study Sponsor (Center for Cancer Research) or their agent(s)

When results of an NIH research study are reported in medical journals or at scientific meetings, the people who take part are not named and identified. In most cases, the NIH will not release any information about your research involvement without your written permission. However, if you sign a release of information form, for example, for an insurance company, the NIH will give the insurance company information from your medical record. This information might

NIH-2977 (4-17)

File in Section 4: Protocol Consent (1)

Version Date: 4/27/2020


affect (either favorably or unfavorably) the willingness of the insurance company to sell you insurance.

If we share your specimens or data with other researchers, in most circumstances we will remove your identifiers before sharing your specimens or data. You should be aware that there is a slight possibility that someone could figure out the information is about you.

Further, the information collected for this study is protected by NIH under a Certificate of Confidentiality and the Privacy Act.

NIH researchers must not share information that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings, for example, if requested by a court.

The Certificate does not protect your information when it:

- 1. is disclosed to people connected with the research, for example, information may be used for auditing or program evaluation internally by the NIH; or
- 2. is required to be disclosed by Federal, State, or local laws, for example, when information must be disclosed to meet the legal requirements of the federal Food and Drug Administration (FDA);
- 3. is for other research;
- 4. is disclosed with your consent.

The Certificate does not prevent you from voluntarily releasing information about yourself or your involvement in this research.

The Certificate will not be used to prevent disclosure to state or local authorities of harm to self or others including, for example, child abuse and neglect, and by signing below you consent to those disclosures. Other permissions for release may be made by signing NIH forms, such as the Notice and Acknowledgement of Information Practices consent.

# **Privacy Act**

The Federal Privacy Act generally protects the confidentiality of your NIH medical information that we collect under the authority of the Public Health Service Act. In some cases, the Privacy Act protections differ from the Certificate of Confidentiality. For example, sometimes the Privacy Act allows release of information from your record without your permission, for example, if it is requested by Congress. Information may also be released for certain research purposes with due consideration and protection, to those engaged by the agency for research purposes, to certain federal and state agencies, for HIV partner notification, for infectious disease or abuse or neglect reporting, to tumor registries, for quality assessment and medical audits, or when the NIH is involved in a lawsuit. However, NIH will only release information from your medical record if it is permitted by both the Certificate of Confidentiality and the Privacy Act.

# **Policy Regarding Research-Related Injuries**

The NIH Clinical Center will provide short-term medical care for any injury resulting from your participation in research here. In general, no long-term medical care or financial compensation for research-related injuries will be provided by the NIH, the NIH Clinical Center, or the Federal

IRB APPROVAL DATE: 06/04/2020

Government. However, you have the right to pursue legal remedy if you believe that your injury justifies such action.

# **Problems or Questions**

If you have any problems or questions about this study, or about your rights as a research participant, or about any research-related injury, contact the Principal Investigator, Christian Hinrichs, MD, <a href="mailto:hinrichs@nih.gov">hinrichs@nih.gov</a>, 240-764-6059. *Other researchers you may call are: Scott Norberg, DO, at 240-858-3303*. You may also call the NIH Clinical Center Patient Representative at 301-496-2626, or the NIH Office of IRB Operations at 301-402-3713, if you have a research-related complaint or concern.

# **Consent Document**

Please keep a copy of this document in case you want to read it again.

| - | read the explanation about this study and questions. I consent to participate in this s | _ |
|---|---|---|
| Signature of Research Participant | Print Name of Research Participa | ant Date |
| explanation about this study and have questions. I am legally authorized to material participant unable to consent and have | LAR) for an Adult Unable to Consents we been given the opportunity to discuss take medical and research decisions on betwee the authority to provide consent to be consent was described to the adult parties study. | ess it and to ask<br>whalf of the adult<br>this study. As |
| Signature of LAR Investigator: | Print Name of LAR | Date |
| Signature of Investigator | Print Name of Investigator | Date |
| | ent process only: This section is only received with a non-English speaking subject a IRB for use as the basis of translation. | |
| Signature of Witness* | Print Name of Witness | Date |

PATIENT IDENTIFICATION

**Consent to Participate in a Clinical Research Study** 

NIH-2977 (4-17) P.A.: 09-25-0099

File in Section 4: Protocol Consent

Version Date: 4/27/2020 IRB NUMBER: 19C0091
 IRB APPROVAL DATE: 06/04/2020

# \*NIH ADMINISTRATIVE SECTION: TO BE COMPLETED BY NIH STAFF IF INTERPRETIVE SUPPORT IS USED. PLEASE CHECK THE BOX THAT APPLIES:

An interpreter, or other individual, who speaks English and the participant's preferred language facilitated the administration of informed consent <u>and served as a witness</u>. The investigator obtaining consent may not also serve as the witness.

An interpreter, or other individual, who speaks English and the participant's preferred language facilitated the administration of informed consent but <u>did not</u> serve as the witness. The name or ID code of the person providing interpretive support is:

PATIENT IDENTIFICATION

Consent to Participate in a Clinical Research Study

NIH-2977 (4-17) P.A.: 09-25-0099

File in Section 4: Protocol Consent

Version Date: 4/27/2020 IRB NUMBER: 19C0091

